CLINICAL TRIAL: NCT03886324
Title: Paclitaxel-Coated Balloon for the Treatment of Symptomatic Recurrent Benign Intestinal Stricture
Brief Title: POISE I Pilot Study
Acronym: POISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GIE Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR2002
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Intestinal Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCB Treatment (Experimental): Stricture patients treated by DCB
  Interventions: Combination Product: GIE Medical Drug Coated Balloon

INTERVENTIONS:
Combination Product: GIE Medical Drug Coated Balloon — Stricture patients treated by DCB

SUMMARY:
POISE I study is a feasibility study for evaluating the safety and efficacy of DCB.

DETAILED DESCRIPTION:
The study is designed to determine the safety and effectiveness for drug coated balloon (DCB) for treating intestinal strictures.

Up to 15 subjects are planned to be enrolled and treated with the study device at up to 5 clinical sites outside of US. Subjects will be followed up post-treatment to one year and then annually for up to 5 years. The annual follow up after the first year is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years.
2. Subjects for whom the balloon dilation would be chosen in standard practice, and the scope could not pass stricture.
3. Recurrent to plain balloon dilation with at least 2 previous balloon dilation or stricturotomy sessions and recurrence of intestine obstructive symptoms/signs.
4. Symptoms of intestinal partial occlusion
5. Length of stenosis/stricture ≤ 7 cm
6. Up to 2 discrete strictures.
7. Ability to undergo periodic endoscopic follow-up.
8. Voluntary participation and provided written informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding or plan to get pregnant in next 12 months.
2. Contraindication to endoscopy, anesthesia or deep sedation.
3. Malignant bowel stricture.
4. Extrinsic benign bowel stricture due to adhesion.
5. Stricture complicated with abscess, fistula, ulceration or associated with mesenteric vessel thrombosis
6. More than 2 stenosis/stricture lesions.
7. Length of stenosis/stricture > 7 cm.
8. Stricture not accessible by endoscopy.
9. Suspected perforation of the gastrointestinal tract
10. Acute bowel obstruction requiring urgent surgical intervention
11. Low rectal or anal strictures
12. Severe coagulation disorders (platelets < 70000; INR > 1.8).
13. Active systemic infection
14. Allergy to paclitaxel or any components of the delivery system.
15. Life expectancy of less than 12 months.
16. Drug abuse or on chronic steroid therapy for comorbidities.
17. Unwilling or unable to comply with the follow-up study requirements.
18. Lacking capacity to provide informed consent.
19. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety.
20. Currently participation in another pre-market drug or medical device clinical study.
21. Chronic steroid use for any medical conditions unless subject is willing to undergo a 4-week washout and discontinue steroid use.
22. Currently requiring abdominal radiation therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incident of serious balloon dilation-related complications | 30 days
  Perforation, bleeding requiring endoscopic or surgical interventions or blood transfusion, severe abdominal pain requiring medications, infection requiring hospitalization or IV antibiotics

SECONDARY OUTCOMES:
Procedure success | 6 months
  defined as subjects who were treated with GIE DCB achieved at least one scale improvement of the Endoscopic Obstructive Scale (EOS).
Percent subjects with improvement in Endoscopic Obstructive Scale (EOS) | 6 months
  Analyzed by 1, 2, or 3 scale improvement.
Change in obstructive symptoms using the Obstructive Symptom Score (OSS). | 30 days, 3 months, 6 months, and 12 months
  The Obstructive Symptom Score (OSS) is a composite measure of the total number of days of obstructive abdominal pain and the severity over a fourteen-day period using a 5-point Likert scale. (1=no pain, 2=mild, 3=moderate, 4=severe, 5=unbearable).
Number of repeated stricture dilation procedures | 30 days, 3 months, 6 months, and 12 months
  Repeat dilation for stricture recurrence
Procedural technical success | Time of procedure
  Successful endoscopic passage followed by successful delivery of the drug-coated balloon to the stricture area without resistance, inflated balloon to the defined diameter, DCB withdraw after deflating balloon without device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Shen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Adventista Hospital, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shen B, Adorno-Garayo CR. Initial safety and efficacy of a novel drug-coated balloon for treatment of benign intestinal strictures. IGIE. 2024 Jan 5;3(1):10-14. doi: 10.1016/j.igie.2023.12.002. eCollection 2024 Mar. PMID 41648897